CLINICAL TRIAL: NCT01592461
Title: START Follow-up Study (NIDA CTN Protocol 0050)
Brief Title: Starting Treatment With Agonist Replacement Therapies Follow-up Study
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Yih-Ing Hser, Professor, University of California, Los Angeles
Other Study IDs: CTN-0050; U10DA013045 (NIH)
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Opioid Dependence
Keywords: Substance abuse treatment outcomes; Opioid dependence; Suboxone; Methadone
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to conduct a follow-up of substance abuse patients (n=1,269) about 2 to 5 years since they were originally recruited from 8 substance abuse treatment clinics (located in 5 states) to participate in a prior clinical trial study called "START" (Starting Treatment with Agonist Replacement Therapies). The START Follow-up Study will be conducted over 5 years and will involve three follow-up interviews with START participants.

The specific aims of the START Follow-up Study are as follows.

1. To determine longer-term outcomes of Suboxone versus methadone treatment received in the START
2. To investigate patient and treatment factors associated with post-START treatment access, utilization, and outcomes among Suboxone and methadone patients
3. To explore other correlates of the long-term outcomes among START patients.

DETAILED DESCRIPTION:
The primary outcome is the trajectory of opioid use since START entry, operationalized as number of days using opioids per month over the follow-up period since START enrollment. Other long-term outcomes of interest will include alcohol and other drug use, mental and physical health, quality of life, criminal justice status, HIV/HCV risk behaviors, and mortality. Treatment access and utilization factors of interest will include: predisposing personal factors, treatment experiences, and perceptions and attitudes toward treatment. Other correlates of interest will include cognitive functioning, mental health functioning, and social support.

2.2 Hypotheses There will be no differences in long-term outcomes of participants randomized to Suboxone treatment versus methadone treatment. To assess this outcome, trajectories of opioid use (operationalized as number of days using opioids per month over the follow-up period since START enrollment) will be analyzed. Other secondary long-term outcomes of interest will also be analyzed and will include alcohol and other drug use, mental and physical health, quality of life, criminal justice status, HIV/HCV risk behaviors, and mortality. Participants with greater access and utilization of treatment, fewer predisposing personal factors, greater social support, and more positive perceptions and attitudes toward treatment, will be more likely to be a member of the low or decreasing drug use trajectories.

2.3 Study Design This longitudinal, observational study will involve contacting the study participants from the original START study for future assessments. The study is expected to be completed in five years.

The follow-up study will consist of three interviews of the START study participants, beginning approximately 2 to 5 years after initial enrollment in the START study and will assess these participants over a 5-year period to provide long-term outcome data 7 to 10 years after START enrollment. This study information will be supplemented by (electronic) medical and other administrative records, as available. An intent-to-treat design will be adopted to include all 1,269 study participants enrolled in START.

Figure 1 presents a summary of the timeline for the conduct of project activities. There will be three participant interviews over the five years of the project. After receiving IRB approval for the conduct of the study, the START community treatment provider (CTP) or Node staff will contact their START participants, obtain participant consent to take part in the follow-up study, and conduct the initial assessment. This assessment will take place in the clinic if possible and by phone if the participant is not able to come in person.

By agreeing to take part in this study the participant will agree to:

1. Updating their locator information initially and throughout the duration of the study;
2. Sharing of clinic and survey data with the lead research team (UCLA);
3. Completing various assessments and providing urine and oral fluid/blood specimens for lab assessments;
4. Providing access to administrative records (e.g., medical records, criminal justice records);
5. Being contacted by the study staff for 2 more interviews in person or by phone (consented prior to each interview).

Local CTP or Node staff will conduct the Visit 1 interview in Years 1-2 of the START follow-up study. Enrollment for the Visit 1 interview will remain open for the life of the study to allow sites that are able to continue to seek participants for Visit 1 beyond Year 2 of the study to do so. The Lead Node staff will conduct the Visit 2 interview by telephone approximately 12 months after the completion of Visit 1. The Lead Node and/or CTP staff will conduct another participant interview approximately 12-18 months after Visit 2 is completed. If a study participant is found late in the study progress for Visit 1, the following visits, 2 and 3 will occur sooner than originally planned, but as far apart as possible. All assessments are completed by the end of Year 5 of the START follow-up study.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate in the study, individuals must have participated in CTN-0027 START.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will include the 1,269 study participants from the original START Study (CTN-0027) that was conducted from 2006 to 2010 at eight community treatment programs (CTPs).
Sampling Method: Non-Probability Sample
Enrollment: 877 (Actual)
Dates: Start 2010-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Opioid use as determined by the Timeline Follow Back measure | from 2006-2009 to 2011-2016
  Opiate use over approximately ten years time period

SECONDARY OUTCOMES:
mortality | from 2006-2009 to 2011-2016
  Rate of mortality over approximately ten years time period

CONTACTS AND LOCATIONS:
Overall Officials: Yih-Ing Hser, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (8):
- United States (8):
  - Matrix Institute on Addictions, Los Angeles, California
  - Bi-Valley Medical Clinic, Inc., Sacramento, California
  - BAART Programs, San Francisco, California
  - Hartford Dispensary, Hartford, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - CODA, Inc., Portland, Oregon
  - NET Steps, Philadelphia, Pennsylvania
  - Evergreen Treatment Services, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared via NIDA Clinical Trials Network Website

REFERENCES:
- [Derived] Hser YI, Zhu Y, Fei Z, Mooney LJ, Evans EA, Kelleghan A, Matthews A, Yoo C, Saxon AJ. Long-term follow-up assessment of opioid use outcomes among individuals with comorbid mental disorders and opioid use disorder treated with buprenorphine or methadone in a randomized clinical trial. Addiction. 2022 Jan;117(1):151-161. doi: 10.1111/add.15594. Epub 2021 Jun 22. PMID 34105213
- [Derived] Evans EA, Yoo C, Huang D, Saxon AJ, Hser YI. Effects of access barriers and medication acceptability on buprenorphine-naloxone treatment utilization over 2 years: Results from a multisite randomized trial of adults with opioid use disorder. J Subst Abuse Treat. 2019 Nov;106:19-28. doi: 10.1016/j.jsat.2019.08.002. Epub 2019 Aug 7. PMID 31540607